CLINICAL TRIAL: NCT01457105
Title: PARTIALLY COVERED NITINOL "ComVi" STENT FOR PALLIATION OF MALIGNANT NON HILAR BILIARY OBSTRUCTION
Brief Title: Covered Self-expandable Metal Stents for Palliation of Malignant Biliary Strictures: Evaluation of a New Type of Stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Professor Guido Costamagna, Professor, Catholic University of the Sacred Heart
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A/1531/05
Record Dates: First submitted 2011-10-19; First posted 2011-10-21 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2011-10

CONDITIONS: Malignant Biliary Strictures
Keywords: Malignant strictures of the main biliary duct

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ComVi biliary stent (Experimental)
  Interventions: Device: Endoscopic retrograde cholangiography (ERC) (ComVi biliary stent)

INTERVENTIONS:
Device: Endoscopic retrograde cholangiography (ERC) (ComVi biliary stent) — Metal stents placement in the main biliary duct during ERC

SUMMARY:
self-expandable metal stents for palliation of malignant biliary strictures

DETAILED DESCRIPTION:
The ComVi biliary stent (Taewoong Medical Inc., Seoul, Korea), is a covered metallic stent with a expanded polytetrafluoroethylene (e-PTFE) membrane sandwiched between two wire layers and has a weaker axial force than other stents.

Patients with middle-distal malignant biliary stricture and with symptoms as jaundice, itching and pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant stenosis at the middle or lower third of the common bile duct inoperable and/or unresectable.
* Patients without liver metastases and 6 months life expectancy
* Patients at the first attempt of endoscopic biliary drainage.
* Negative history for biliary tract surgery.

Exclusion Criteria:

* Patients with ampullary cancer.
* Patients with hilar and/or intra-hepatic ducts malignancy.
* Patients with haemobilia.
* Patients with acute cholangitis at the time of stenting.
* Patients with previous percutaneous, endoscopic or surgical biliary drainage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
patency and effectiveness of the ComVi stent in palliation of jaundice in patients with malignant biliary strictures | two years

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University, Rome, RM, Italy